CLINICAL TRIAL: NCT06565754
Title: Effect of Adding Blood Flow Restriction to Strengthening Exercise in Patients With Patellofemoral Pain Syndrome
Acronym: BFR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Mahmoud Abdelaziz Khalil, doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P.T.REC/012/005148; P.T.REC/012/005148 (Other: ethical committee faculty of physical therapy CU)
Record Dates: First submitted 2024-07-26; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: BFR; PFPS; Strengthening Exercises; Quadriceps Strength; Dynamic Balance; Joint Position Sense
Keywords: PFPS; Patellofemoral Pain Syndrome; Blood Flow Restriction Training; Strengthening Exercises; Dynamic Balance
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- strengthening exercises group (SE Group) (Active Comparator): all patients will receive :
  1. Isometric quadriceps exercise - 3 sets of 20 repetitions (5 s).
  2. Straight leg raise (SLR) with 3 sets - 20 repetitions.
  3. Short arc knee extension exercise - 3 sets of 20 repetitions.
  4. Hip abduction from side lying - 3 sets of 20 repetitions.
  Interventions: Other: strengthening exercise
- BFRT plus strengthening exercises group (BFRT Group) (Experimental): all patients will receive the below exercises using BFR cuff :
  1. Isometric quadriceps exercise - 3 sets of 20 repetitions (5 s).
  2. Straight leg raise (SLR) with 3 sets - 20 repetitions.
  3. Short arc knee extension exercise - 3 sets of 20 repetitions.
  4. Hip abduction from side lying - 3 sets of 20 repetitions.
  Interventions: Other: BFR; Other: strengthening exercise

INTERVENTIONS:
Other: BFR — Blood flow restriction training is an accessory to a variety of different exercise modes (e.g., resistance exercise, walking, cycling) has recently become a popular research topic. It involves the application of pressurized cuffs to the proximal portion of each lower extremity or upper extremity. It enhance blood pooling in the capillary beds of the limb muscles distal to the tourniquet or cuff.
  The 3rd Generation SmartCuffs® pump (SmartCuffs® 3.0 PRO) is Personalized Pressure feature which allows for a fast, hassle-free personalized pressure calculation. With the built-in pressure sensor and on-board computer, it is calculate arterial occlusion pressure and set the optimal pressure for patient's body. There is no need for an external doppler probe or hand pump. This unit will do everything for patient. Smart Cuffs 3rd generation is FDA Approved Listed Class 1 device.
  The automatized tourniquet (Smart Tools) contains a ring-shaped single- chamber
  Arms: BFRT plus strengthening exercises group (BFRT Group)
Other: strengthening exercise — Quadriceps strengthening exercises are part of the treatment of PFPS, but the heavy resistance exercises may aggravate knee pain. Blood flow restriction training (BFRT) provides a low-load quadriceps strengthening method to treat PFPS (Giles et al., 2017).

SUMMARY:
To study the effect of adding BFRT to strengthening exercises and compare it with strengthening exercises alone in improving, muscular strength, pain, function, joint position sense, and dynamic balance test (star excursion test). in patients with PFPS.

DETAILED DESCRIPTION:
Background: Patellofemoral Pain Syndrome (PFPS) is a common condition characterized by anterior knee pain, particularly affecting individuals aged 15-30. It often involves lower limb muscle weakness, particularly in the quadriceps, which can exacerbate symptoms and affect functional performance. Blood Flow Restriction Training (BFRT) has shown promise in enhancing muscle strength and functional outcomes with reduced intensity compared to traditional high-intensity training.

Purpose: This study aims to compare the efficacy of combining BFRT with traditional strengthening exercises versus using strengthening exercises alone in improving muscular strength, pain, function, joint position sense, and dynamic balance in patients with PFPS.

Methods: A triple-blinded, randomized controlled trial was conducted at the Almenshawy General Hospital, Tanta, Egypt. Fifty patients with unilateral non-traumatic PFPS, aged 18-35, were randomly assigned to either a strengthening exercises group (SE Group) or a BFRT plus strengthening exercises group (BFRT Group). Both groups underwent a 6-week intervention with three sessions per week. Outcomes assessed included quadriceps and hip abductors strength, pain severity (Visual Analog Scale), functional status (Kujala Patellofemoral Score), joint position sense (measured by digital inclinometer), and dynamic balance (Star Excursion Balance Test).

ELIGIBILITY:
Inclusion Criteria:

* Patient referred from Orthopedic surgeon with diagnosis of patellofemoral pain syndrome PFPS.
* Both genders.
* BMI ranges from 18.5 to 29.9.
* Age ranges between 18 and 40 years experienced non-traumatic PFPS onset of anterior knee pain for greater than 2 weeks.
* Pain with any two activities, including running, jumping, squatting, kneeling, stair ascent/descent or prolonged sitting.

Exclusion Criteria:

* Coexisting pathology around the knee, including patellar subluxation or dislocation.
* Other sources of anterior knee pain (bursa, fat pad).
* Previous knee surgery.
* Suspicion of patellar tendinopathy, with strong consideration of pain localised to the patellar tendon.
* Any cardiovascular disease.
* Uncontrolled hypertension.
* Any lower limb trauma.
* Hip and ankle pathology.
* BMI more than 30%.
* Pregnancy.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
quadriceps and hip abductors strength | 6 weeks
  Hand-Held Dynamometer (HHD). The Lafayette® HHD is a valid and reliable instrument of low cost and easy handling compared to the isokinetic dynamometer for assessment of muscle strength

SECONDARY OUTCOMES:
pain severity using Visual Analog Scale (VAS) | 6 weeks
  The Visual Analog Scale is determined by measuring in millimeters from the left end of the line to the patient's mark. Participants will ask to determine the point at which pain represents the severity of pain maximum is 10 while lowest level of pain is zero
functional status (Kujala Patellofemoral Score) | 6 weeks
  The 13 items on the scale are used to assess subjective symptoms and functional restrictions. A score can have a minimum of 0 points or a maximum of 100 points.
joint position sense (measured by digital inclinometer) | 6 weeks
  Digital Inclinometer for joint position sense assessment. Device (Digital Protractor, 82201b-00, INSPEC, China) The inclinometer is a valid and reliable method to assess the knee proprioception through JPS in open kinetic chain
dynamic balance (Star Excursion Balance Test | 6 weeks
  Four strips of adhesive tape will need to be cut to a length of 6-8 feet each. Two pieces will be used to form a '+', with the other two being placed over top to form an 'x' so that a star shape is formed. It is important that all lines are separated from each other by a 45° angle. The goal of the Star Excursion Balance Test (SEBT) is to maintain single leg stance on one leg while reaching as far as possible with the contralateral leg.

CONTACTS AND LOCATIONS:
Overall Officials: enas F youssef, Professor, Study Chair — Cairo University; abdelgalil A shaaban, PhD, Study Director — Cairo University; ahmed S helal, PhD, Study Director — Tanta University; ahmed M khalil, PhD, Study Director — Pharos University in Alexandria
Locations (1):
- Cairo University, Giza, Egypt

REFERENCES:
- [Background] Stefanov F, Morris L, Elhelali A, Kavanagh EP, Lundon V, Hynes N, Sultan S. Insights from complex aortic surgery with a Streamliner device for aortic arch repair (STAR). J Thorac Cardiovasc Surg. 2016 Nov;152(5):1309-1318.e5. doi: 10.1016/j.jtcvs.2016.06.043. Epub 2016 Jun 29. PMID 27485677
- [Background] Sigaud O, Stulp F. Policy search in continuous action domains: An overview. Neural Netw. 2019 May;113:28-40. doi: 10.1016/j.neunet.2019.01.011. Epub 2019 Feb 5. PMID 30780043
- [Background] Golbs A, Nimmervoll B, Sun JJ, Sava IE, Luhmann HJ. Control of programmed cell death by distinct electrical activity patterns. Cereb Cortex. 2011 May;21(5):1192-202. doi: 10.1093/cercor/bhq200. Epub 2010 Oct 21. PMID 20966045
- [Background] Panneton WM, Gan Q, Juric R. The rat: a laboratory model for studies of the diving response. J Appl Physiol (1985). 2010 Apr;108(4):811-20. doi: 10.1152/japplphysiol.00600.2009. Epub 2010 Jan 21. PMID 20093670
- [Background] Wang H, Li Y, Zhang C, Han Y, Zhang X, Zhu T, Li T. Immunological and virological responses to cART in HIV/HBV co-infected patients from a multicenter cohort. AIDS. 2012 Sep 10;26(14):1755-63. doi: 10.1097/QAD.0b013e328355ced2. PMID 22614885
- [Background] Zhang A, Mo X, Zhou N, Wang Y, Wei G, Chen J, Chen K, Ouyang P. A novel bacterial beta-N-acetyl glucosaminidase from Chitinolyticbacter meiyuanensis possessing transglycosylation and reverse hydrolysis activities. Biotechnol Biofuels. 2020 Jun 29;13:115. doi: 10.1186/s13068-020-01754-4. eCollection 2020. PMID 32612678
- [Background] Ziegler MG, Milic M, Lu X, Gharaibeh M, Elayan H. Effect of obstructive sleep apnea on the response to hypertension therapy. Clin Exp Hypertens. 2017;39(5):409-415. doi: 10.1080/10641963.2016.1259327. Epub 2017 May 30. PMID 28557555
- [Background] Herzog N, Hartkamp JD, Verheugd P, Treude F, Forst AH, Feijs KL, Lippok BE, Kremmer E, Kleine H, Luscher B. Caspase-dependent cleavage of the mono-ADP-ribosyltransferase ARTD10 interferes with its pro-apoptotic function. FEBS J. 2013 Mar;280(5):1330-43. doi: 10.1111/febs.12124. Epub 2013 Feb 13. PMID 23305266
- [Background] Barrett CL, Mann GE, Taylor PN, Strike P. A randomized trial to investigate the effects of functional electrical stimulation and therapeutic exercise on walking performance for people with multiple sclerosis. Mult Scler. 2009 Apr;15(4):493-504. doi: 10.1177/1352458508101320. Epub 2009 Mar 12. PMID 19282417
- [Background] Parnia S, Yang J, Nguyen R, Ahn A, Zhu J, Inigo-Santiago L, Nasir A, Golder K, Ravishankar S, Bartlett P, Xu J, Pogson D, Cooke S, Walker C, Spearpoint K, Kitson D, Melody T, Chilwan M, Schoenfeld E, Richman P, Mills B, Wichtendahl N, Nolan J, Singer A, Brett S, Perkins GD, Deakin CD. Cerebral Oximetry During Cardiac Arrest: A Multicenter Study of Neurologic Outcomes and Survival. Crit Care Med. 2016 Sep;44(9):1663-74. doi: 10.1097/CCM.0000000000001723. PMID 27071068
- [Background] Galvez-Martinez S, Mateo-Marti E. Ultraviolet Irradiation on a Pyrite Surface Improves Triglycine Adsorption. Life (Basel). 2018 Oct 25;8(4):50. doi: 10.3390/life8040050. PMID 30366364
- [Background] Saade Riachy C, Nemr E. Medical professionalism in Lebanon: between doctors' perception and patients' satisfaction. Int J Med Educ. 2020 Aug 21;11:171-172. doi: 10.5116/ijme.5f28.77a3. No abstract available. PMID 32827248
- [Background] Maher SK, Wojnarowicz P, Ichu TA, Veldhoen N, Lu L, Lesperance M, Propper CR, Helbing CC. Rethinking the biological relationships of the thyroid hormones, l-thyroxine and 3,5,3'-triiodothyronine. Comp Biochem Physiol Part D Genomics Proteomics. 2016 Jun;18:44-53. doi: 10.1016/j.cbd.2016.04.002. Epub 2016 Apr 7. PMID 27085304
- [Background] Ozbay B, Uzun K, Arslan H, Zehir I. Functional and radiological impairment in women highly exposed to indoor biomass fuels. Respirology. 2001 Sep;6(3):255-8. doi: 10.1046/j.1440-1843.2001.00339.x. PMID 11555385
- [Background] Martelletti P, Schwedt TJ, Lanteri-Minet M, Quintana R, Carboni V, Diener HC, Ruiz de la Torre E, Craven A, Rasmussen AV, Evans S, Laflamme AK, Fink R, Walsh D, Dumas P, Vo P. My Migraine Voice survey: a global study of disease burden among individuals with migraine for whom preventive treatments have failed. J Headache Pain. 2018 Nov 27;19(1):115. doi: 10.1186/s10194-018-0946-z. PMID 30482181
- [Background] Esparza Martin N. [Hypotonic hiponatremia. Differential diagnosis]. Med Clin (Barc). 2016 Dec 2;147(11):507-510. doi: 10.1016/j.medcli.2016.09.013. Epub 2016 Oct 27. No abstract available. Spanish. PMID 28126145
- [Background] Jagadeesh AT, Puttur A, Mondal S, Ibrahim S, Udupi A, Prasanna LC, Kamath A. Devising focused strategies to improve organ donor registrations: A cross-sectional study among professional drivers in coastal South India. PLoS One. 2018 Dec 21;13(12):e0209686. doi: 10.1371/journal.pone.0209686. eCollection 2018. PMID 30576381
- [Background] Huijbers MG, Querol LA, Niks EH, Plomp JJ, van der Maarel SM, Graus F, Dalmau J, Illa I, Verschuuren JJ. The expanding field of IgG4-mediated neurological autoimmune disorders. Eur J Neurol. 2015 Aug;22(8):1151-61. doi: 10.1111/ene.12758. Epub 2015 May 29. PMID 26032110
- [Background] Selak V, Webster R, Stepien S, Bullen C, Patel A, Thom S, Arroll B, Bots ML, Brown A, Crengle S, Dorairaj P, Elley CR, Grobbee DE, Harwood M, Hillis GS, Laba TL, Neal B, Peiris D, Rafter N, Reid C, Stanton A, Tonkin A, Usherwood T, Wadham A, Rodgers A. Reaching cardiovascular prevention guideline targets with a polypill-based approach: a meta-analysis of randomised clinical trials. Heart. 2019 Jan;105(1):42-48. doi: 10.1136/heartjnl-2018-313108. Epub 2018 Jun 28. PMID 29954855
- [Background] Muoio R, Caretti C, Rossi L, Santianni D, Lubello C. Letter to the Editor: Water safety plans and risk assessment: A novel procedure applied to treated water turbidity and gastrointestinal diseases. Int J Hyg Environ Health. 2020 Aug;229:113455. doi: 10.1016/j.ijheh.2020.113455. Epub 2020 Jan 25. No abstract available. PMID 31992522
- [Background] Nakao S, Platek A, Hirano S, Takeichi M. Contact-dependent promotion of cell migration by the OL-protocadherin-Nap1 interaction. J Cell Biol. 2008 Jul 28;182(2):395-410. doi: 10.1083/jcb.200802069. Epub 2008 Jul 21. PMID 18644894
- [Background] Kasten P, Pape G, Raiss P, Bruckner T, Rickert M, Zeifang F, Loew M. Mid-term survivorship analysis of a shoulder replacement with a keeled glenoid and a modern cementing technique. J Bone Joint Surg Br. 2010 Mar;92(3):387-92. doi: 10.1302/0301-620X.92B3.23073. PMID 20190310
- [Background] Froon-Torenstra D, Beket E, Khader AM, Hababeh M, Nasir A, Seita A, Benninga MA, van den Berg MM. Prevalence of functional constipation among Palestinian preschool children and the relation to stressful life events. PLoS One. 2018 Dec 6;13(12):e0208571. doi: 10.1371/journal.pone.0208571. eCollection 2018. PMID 30521620
- [Background] Abe T, Kearns CF, Sato Y. Muscle size and strength are increased following walk training with restricted venous blood flow from the leg muscle, Kaatsu-walk training. J Appl Physiol (1985). 2006 May;100(5):1460-6. doi: 10.1152/japplphysiol.01267.2005. Epub 2005 Dec 8. PMID 16339340
- [Background] Abe T, Fujita S, Nakajima T, Sakamaki M, Ozaki H, Ogasawara R, Sugaya M, Kudo M, Kurano M, Yasuda T, Sato Y, Ohshima H, Mukai C, Ishii N. Effects of Low-Intensity Cycle Training with Restricted Leg Blood Flow on Thigh Muscle Volume and VO2MAX in Young Men. J Sports Sci Med. 2010 Sep 1;9(3):452-8. eCollection 2010. PMID 24149640
- [Background] Abbas MJ, Dancy ME, Marigi EM, Khalil LS, Jildeh TR, Buckley PJ, Gillett J, Burgos W, Okoroha KR. An Automated Technique for the Measurement of Limb Occlusion Pressure During Blood Flow Restriction Therapy Is Equivalent to Previous Gold Standard. Arthrosc Sports Med Rehabil. 2022 May 28;4(3):e1127-e1132. doi: 10.1016/j.asmr.2022.04.002. eCollection 2022 Jun. PMID 35747637
- [Result] Penailillo L, Blazevich AJ, Nosaka K. Factors contributing to lower metabolic demand of eccentric compared with concentric cycling. J Appl Physiol (1985). 2017 Oct 1;123(4):884-893. doi: 10.1152/japplphysiol.00536.2016. Epub 2017 Jun 29. PMID 28663378
- See also: This review found that BFR significantly improves muscle strength but is less effective than heavy-load training . BFR is a viable and tolerable rehab tool, needing personalized — https://bjsm.bmj.com/content/51/13/1003.abstract
- See also: The study examines how low-intensity cycling with and without blood flow restriction (BFR) impacts muscle strength, hypertrophy, and aerobic capacity, addressing whether BFR can simultaneously enhance both muscular and cardiovascular fitness. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3761718/
- Available data/document: Study Protocol — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10563562/